CLINICAL TRIAL: NCT01368575
Title: The Effect of Different Surgical Methods in the Treatment of Patients With Ischemic Mitral Regurgitation and Assess the Dynamics of Heart Failure and the Effectiveness of Surgical Treatment of Mitral Valve.
Brief Title: Surgical Treatment of Ischemic Mitral Regurgitation
Acronym: TIME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIME-002
Record Dates: First submitted 2011-05-24; First posted 2011-06-08 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Mitral Valve Insufficiency
Keywords: Ischemic; Mitral; Valve; Insufficiency; SVR
MeSH Terms: conditions — Mitral Valve Insufficiency; Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- subgroup B1 (Active Comparator): subgroup B1 will receive CABG combined with MV repair with annuloplasty rigid ring
  Interventions: Procedure: CABG combined with MV repair with remodeling annuloplasty rigid ring
- subgroup B2 (Active Comparator): B2 - CABG combined with MV repair with remodeling annuloplasty rigid ring and endoventricularplasty of subvalvular apparatus
  Interventions: Procedure: CABG combined with MV repair with remodeling annuloplasty rigid ring and endoventricularplasty of subvalvular apparatus
- subgroup A2 (Active Comparator): CABG combined with MV repair with remodeling annuloplasty rigid ring
  Interventions: Procedure: CABG combined with MV repair with remodeling annuloplasty rigid ring
- subgroup A1 (Active Comparator): only CABG
  Interventions: Procedure: CABG
- subgroup B3 (Active Comparator): patients in subgroup B3 will be performed CABG and MV replacement with preservation of subvalvular apparatus
  Interventions: Procedure: CABG and MV replacement

INTERVENTIONS:
Procedure: CABG — CABG
  Other Names: will be performed only CABG (subgroup A1)
  Arms: subgroup A1
Procedure: CABG combined with MV repair with remodeling annuloplasty rigid ring — CABG combined with MV repair with remodeling annuloplasty rigid ring
  Arms: subgroup A2
Procedure: CABG combined with MV repair with remodeling annuloplasty rigid ring — CABG combined with MV repair with remodeling annuloplasty rigid ring
  Other Names: patients in subgroup B1 will receive CABG combined with MV repair with remodeling annuloplasty rigid ring
  Arms: subgroup B1
Procedure: CABG combined with MV repair with remodeling annuloplasty rigid ring and endoventricularplasty of subvalvular apparatus — CABG combined with MV repair with remodeling annuloplasty
  Other Names: CABG grafting combined with MV repair with remodeling annuloplasty and endoventricularplasty of subvalvular
  Arms: subgroup B2
Procedure: CABG and MV replacement — coronary artery bypass grafting and mitral valve replacement
  Other Names: patients in subgroup B3 will be performed CABG and MV replacement with preservation of subvalvular apparatus
  Arms: subgroup B3

SUMMARY:
The primary objective is to estimate surgical treatment (prosthesis or plastic) of moderate and severe ischemic mitral regurgitation combined with CABG in patients with CAD and impact on heart failure and progress of mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female between 30 to 75 years of age (inclusive) on the day of signing the informed consent.
* Patients with a verified diagnosis of CAD, including post myocardial infarction scar.
* Coronary artery pathology to be coronary artery bypasses grafting.
* The presence of moderate or severe ischemic mitral regurgitation.

Exclusion Criteria:

* The patient did not sign the informed consent.
* Aortic valve disease requiring prosthetic or aortic valve repair.
* Organic lesion of valve and subvalvular structures (endocarditis and degenerative processes of the mitral valve).

  а) separation of the mitral valve chords; б) rupture and perforation of the mitral valve; в) myxomatous degeneration and calcification of the mitral valve
* Patients with acute coronary syndrome.
* The presence of the indications for angioplasty of the coronary arteries.
* Coronary artery bypasses grafting in history.
* Parallel patient participation in other studies.
* The organs diseases, which can be reason to death after surgery during the first 3 years.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Assess the degree of mitral regurgitation in the early and late term of the study. Identify the cause of the return of IMR. Determine the dynamics of heart failure in patients with IMR. | 3,6,12,24,36 months

SECONDARY OUTCOMES:
Assessment of IMR | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Cherniavskiy, MD, PhD, Principal Investigator — State Research Institute of Circulation Patholody Novosibirsk, 630055 Russian Federation
Locations (1):
- State Research Institute of Circulation Patholody, Novosibirsk, Russia